CLINICAL TRIAL: NCT01353534
Title: A Phase 1/2, Randomized, Open-Label, Study to Assess the Immunogenicity and Safety of a Vaccine Enhancement Patch (VEP) When Administered With Two Doses of Intramuscular Inactivated Influenza H5N1 Vaccine in Healthy Adults
Brief Title: Open-label Study to Assess Immunogenicity and Safety of a Vaccine Enhancement Patch When Administered With 2 Doses of H5N1 Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC82-102
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Immunogenicity and Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 3.8 mcg with AS03 adjuvant at D0 and 21
  Interventions: Biological: A/H5N1 Antigen
- Group 2 (Experimental): 15 mcg at D0 and 21
  Interventions: Biological: A/H5N1 Antigen
- Group 3 (Experimental): 15 mcg + 50 mcg VEP at D0 and 21
  Interventions: Biological: A/H5N1 Antigen; Drug: Vaccine Enhancement Patch
- Group 4 (Experimental): 30 mcg + 50 mcg VEP at D0
  Interventions: Biological: A/H5N1 Antigen; Drug: Vaccine Enhancement Patch

INTERVENTIONS:
Biological: A/H5N1 Antigen — A/H5N1 Antigen
Drug: Vaccine Enhancement Patch — Vaccine Enhancement Patch
  Arms: Group 3; Group 4

SUMMARY:
Groups 1 to 3 will receive two vaccinations on Day 0 and Day 21. Group 1 will receive 3.8µg A/H5N1 antigen formulated with AS03 adjuvant, administered by IM injection. Group 2 will receive 15µg A/H5N1 by IM alone. Group 3 will also receive 15µg A/H5N1 antigen administered IM but followed by the topical application of a VEP at the vaccination site. Group 4 will receive a single vaccination on Day 0 of 30µg A/H5N1antigen by IM, followed by application of a VEP at the vaccination site.

The VEP (Vaccine Enhancement Patch) contains 50 mcg LT (heat-labile enterotoxin of E. coli)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females 18-49 years of age (inclusive)
* signed Informed Consent
* Women who are not post-menopausal or surgically sterile must have a negative serum or urine pregnancy test at screening and at all in-clinic visits with understanding to not become pregnant over the duration of the study.

Exclusion Criteria:

* Clinically significant laboratory abnormalities at screening
* abnormalities at physical examination
* known allergies to any component of the A/H5N1 antigen
* known egg protein allergy
* known allergies to adhesives
* known coagulation disorders
* use of any anticoagulant medication within 30 days prior to vaccination or planned usage during the study period
* participated in research involving investigational product within 30 days before planned date of vaccination or planned participation during study period
* donated or received blood or blood products such as plasma within the three months before planned date of vaccination or planned donation or use during the study period
* received or planned receipt of seasonal influenza vaccine during the study period
* received any licensed vaccines within 2 weeks (inactivated vaccines) or 4 weeks (live vaccines) prior to planned date of vaccination
* planned receipt of any licensed vaccine during the first 42 days on study
* previous or planned vaccination with any vaccine containing an oil in water emulsion adjuvant
* previous or planned vaccination with pandemic vaccine against A/H5N1 or previous proven contact with A/H5N1 wild type virus
* ever received investigational enterotoxigenic E. coli LT, or LT (R192G) or NasalFlu, Berna Biotech, Ltd. Ever received cholera toxin or vaccine
* Recent or regular use of oral, topical or injected steroid medications within 30 days prior to vaccination or planned use during the study period.
* Use of immunosuppressive systemic steroid medications including inhaled steroids within three months prior to vaccination or planned use during the study period
* Comorbid conditions or treatments that are immunosuppressive, including cancer, diabetes, and end-stage renal disease, as determined by the Investigator
* positive serology for HIV-1, HIV-2, HBsAg, or HCV
* history of severe atopy
* medical history of acute or chronic skin disease at vaccination area
* active skin allergy
* signs of acute skin infection, sunburn or skin abnormalities at the vaccination area including fungal infections, severe acne, active contact dermatitis, or a history of keloid formation
* hirsute at vaccination area
* artificial tanning over the duration of the study including the screening period
* visible tattoos or marks at the vaccination area that would prevent appropriate dermatologic monitoring of the vaccination site
* fever greater than or equal to 38.0°C at the time of planned vaccination
* suspicion of or recent history of alcohol or substance abuse
* women who are pregnant or breastfeeding
* acute illness at screening or at the time of planned vaccination
* ever had a serious reaction to prior influenza vaccination
* developed a neurological disorder following a previous influenza vaccination or have any acute and evolving neurological disorder
* employee of the investigational site or sponsor
* history of employment in bird or poultry industries or considerable exposure to birds

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluate hemagglutination inhibition (HI) immune responses | Day 42
  Evaluate hemagglutination inhibition (HI) immune responses to two doses of 15μg A/H5N1 achieved in the antigen plus VEP group versus the antigen alone group (Group 3 vs. Group 2) at Day 42 using standard serological parameters (Geometric Mean Titer [GMT], Geometric Mean Fold Ratio [GMFR], seroconversion and seroprotection).

SECONDARY OUTCOMES:
Safety of 15µg and 30µg IM A/H5N1 antigen administered with the 50µg VEP | 8 months
  Comprehensive assessment of solicited and non-solicited local (vaccination site) and systemic adverse events (AEs) Safety follow-up through six months after last vaccination
Characterize HI immune responses | 8 months
  Characterize HI immune responses in the 15µg A/H5N1 antigen alone group (Group 2) and the 15µg A/H5N1 antigen plus VEP group (Group 3) to determine if levels meet or exceed EMA CPMP/BWP/214/96 criteria for immunogenicity:
  * The percent of subjects achieving seroconversion for HI antibody titer should meet or exceed 40%
  * The percent of subjects achieving an HI antibody titer ≥ 1:40 should meet or exceed 70%
  * GMT increase > 2.5

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, MD, Principal Investigator — Medical University of Vienna
Locations (5):
- Austria (3):
  - Privatklinik Leech, Graz, Graz
  - Medizinische Universität Wien, Vienna, Vienna
  - Medical University of Vienna, Vienna
- Belgium (2):
  - Antwerp University - Campus Drie Eiken, Antwerp, Antwerp
  - University Hospital Ghent, Ghent, Ghent